CLINICAL TRIAL: NCT05555758
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics Profile of Aom0319 in Healthy White Subjects
Brief Title: Aom0319 SAD Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amckaus PTY LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aom0319-ACT-01
Record Dates: First submitted 2022-09-19; First posted 2022-09-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): Four ascending dose levels of Aom0319 (n=24) for intravenous injection for once. Dosage day is Day 1.
  Interventions: Drug: Adamgammadex Sodium
- placebo group (Placebo Comparator): Four ascending dose levels of placebo (n=8) for intravenous injection for once. Dosage day is Day 1.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Adamgammadex Sodium — Aom0319 will be administered intravenously with water for injection.
  Other Names: Aom0319
  Arms: experimental group
Drug: 0.9% Sodium Chloride Injection — 0.9% Sodium Chloride will be administered intravenously.
  Other Names: Placebo
  Arms: placebo group

SUMMARY:
Only SAD study will be conducted in this project. SAD represents single ascending dose. Multiple ascending dose have been cancelled. This decision has been made at the discretion of the Sponsor.

DETAILED DESCRIPTION:
This study was designed to evaluate the safety and tolerability of Aom0319.

The trial is designed as follows.

1. SAD: 32 participants will be studied in four groups with n = 8 (6 active: 2 placebo) per group.

ELIGIBILITY:
Inclusion Criteria

1. Healthy male or female subjects ≥18 years and ≤55 years of age on the day of ICF signing.
2. Subjects must be White (participants from Europe, Middle East, North Africa, Australia, and New Zealand are permitted), with biological parents and both sets of biological grandparents also be White;
3. Male subjects must have a body weight ≥50 kg and female subjects must have a body weight ≥45 kg. Body mass index (calculated as weight [kg]/height [m]2) must be ≥18.0 and ≤ 32.0 kg/m2;
4. In good health, as determined by medical history, physical examination, clinical laboratory evaluation, 12-lead ECG, and vital signs (including oxygen saturation) within normal range or deemed by the investigator to be not clinically significant;
5. Willing to use an adequate method of contraception, and do not plan to become pregnant, impregnate a partner, or donate sperm or ova throughout the study and for 3 months following the end of the study. Abstinence is an acceptable method of contraception provided it aligns with the preferred and usual lifestyle of the subject. Female subjects of nonchildbearing potential and subjects who are exclusively in same-sex relationships are exempt from contraception requirements. An adequate method of contraception is defined as:

   a)For female subjects, an adequate method of contraception is defined as the use of a condom by the male partner combined with the use of a highly effective method of contraception. The following are considered as highly effective methods of contraception: i)A nonhormonal intrauterine device; ii)Bilateral tubal occlusion (e.g. Essure-non-surgical sterility procedure and Bilateral tubal ligation), and/or a vasectomized partner with documented azoospermia 90 days after procedure, if that partner is the sole sexual partner; b)For male subjects, an adequate method of contraception is defined as use of a condom combined with the use of a highly effective method of contraception by the female partner of childbearing potential. A highly effective method of contraception is i)Oral contraceptives containing combined estrogen and progesterone, a vaginal ring, injectable and implantable hormonal contraceptives, intrauterine hormone-releasing system (e.g. Mirena) and progestogen-only hormonal contraception associated with inhibition of ovulation; ii)A hormonal or nonhormonal intrauterine device; iii)Bilateral tubal occlusion including bilateral tubal ligation, and/or a vasectomized subject with documented azoospermia 90 days after procedure, if that partner is the sole sexual partner;
6. Female subjects must be non-pregnant (confirmed by a negative serum [at screening] and urine [on Day -1] pregnancy test), non-lactating, or be of nonchildbearing potential (females who have been postmenopausal [defined as 12 months of amenorrhea in the absence of other biological cause with confirmatory follicle stimulating hormone ≥40 IU/L] for at least 12 consecutive months or are surgically sterile [hysterectomy or bilateral oophorectomy or bilateral complete salpingectomy]);
7. Willing and able to freely given informed consent by signing the ICF.

Exclusion Criteria:

1. History of hereditary bleeding disorders, coagulation disorders, non-traumatic bleeding requiring treatment, or thromboembolism; or currently have any disease that can cause bleeding (including coagulation disorder, thrombocytopenia [platelet count < 150×109/L] and prothrombin time-international normalized ratio >1.5);
2. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥1.5 × the upper limit of normal at screening or check-in;
3. Abnormal ECG results which are judged as clinically significant by the investigator, or any of the following:

   1. QTcF interval (calculated as QTc=QT/[RR^0.33]) >430 ms for male subjects and > 450 ms for female subjects;
   2. Complete bundle branch block including left and/or right complete bundle branch block;
   3. Symptoms of acute or age variable myocardial infarction;
   4. ST-T changes suggestive of myocardial ischemia;
   5. First-degree (PR interval ≥200 ms), second-degree, or third-degree atrioventricular block;
4. Abnormal blood pressure or heart rate (defined as systolic blood pressure >140 mmHg or <90 mmHg, diastolic blood pressure >90 mmHg or <50 mmHg, and heart rate <45 bpm or >100 bpm) during the study screening period and at check-in;
5. Febrile illness or infection within 7 days prior to drug administration (Day 1);
6. History of significant food or drug allergy or allergy history (including symptoms of allergic reaction, clinically significant skin diseases such as contact dermatitis or psoriasis, visible skin rashes, or asthma attacks during physical examination) which is judged as clinically significant by the investigator, or hypersensitivity to cyclodextrin;
7. Subjects who have previously taken sugammadex sodium;
8. Acute or chronic clinically significant infectious disease during the screening period or at check-in; or a positive hepatitis C antibody, human immunodeficiency virus antibody, hepatitis B surface antigen, or reactive HIV antigen/antibody at screening;
9. History or manifestation of disease that, in the opinion of the investigator, renders the subject unsuitable for the study, including but not limited to nervous system, cardiovascular, blood, lymphatic, immune, kidney, liver, gastrointestinal, respiratory, metabolic, and musculoskeletal disorders;
10. History of tuberculosis (TB) or related infection that is active, latent, or inadequately treated, or positive TB test (QuantiFERON Gold);
11. History of disseminated herpes zoster, disseminated herpes simplex, recurrent localized cutaneous herpes zoster (including one episode of cutaneous herpes zoster);
12. Poor peripheral venous access, unable to tolerate venipuncture, or have a significant history of trypanaphobia or hemophobia;
13. History of substance abuse (including illicit drugs) within 6 months prior to dosing (Day 1);
14. Use of drugs of abuse (including but not limited to amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxy-methamphetamine, phencyclidine, and tetrahydrocannabinol) within 3 months prior to dosing (Day 1), or positive drugs of abuse test at screening or Day -1;
15. Those who have been dosed in a previous study or administration of an investigational drug within 1 month (or 5 half-lives, whichever is longer) prior to dosing (Day 1);
16. Use of fusidic acid, toremifene citrate, tamoxifen citrate, clomiphene citrate, progesterone, norethisterone, testosterone, prednisone, combination contraceptives that contain steroid hormones such as progesterone, other steroid hormones, which could affect the absorption or PK parameters of Aom0319 within 7 days prior to dosing (Day 1) until discharge;
17. Donation or loss of blood exceeding 500 mL of blood within 56 days prior to dosing (Day 1), plan to donate blood or blood components during the study period, or have previously received blood products;
18. With the exception of those listed in exclusion criterion #16, use of prescription drugs, over-the-counter drugs, Chinese herbal medicines, dietary supplements, or natural health products (including vitamins, minerals, and phytotherapeutic, herbal, and plant-derived preparations) from 2 weeks prior to dosing (Day 1) until discharge;
19. Administration of a vaccine within 4 weeks prior to dosing (Day 1) or plan to be vaccinated during the study;
20. Smoke more than 5 cigarettes per day within 30 days prior to dosing (Day 1) or inability to abstain from tobacco- or nicotine-containing products during the study (from Day -1 to the follow up visit);
21. Regular consumption of the amount of alcohol (in an Australian standard drink）of more than 2 standard drinks per day or 14 standard drinks per week within 3 months prior to check-in (Day -1; 1 standard drink is equivalent to 10 grams of alcohol: approximately 285 mL full-strength beer or cider[4.9% alc/vol], 375 ml mid-strength beer[3.5% alc/vol], 425ml light- strength beer[2.7% alc/vol], 100 mL wine or 30 mL shot of 40% spirit ). A positive alcohol breath test at screening or check-in (Day -1), or inability to abstain from alcohol during the study from check-in (Day -1) to the follow-up visit;
22. Daily regular consumption of tea, coffee, and/or caffeinated beverages exceeding 8 cups (where 1 cup = 250 mL) within 3 months prior to dosing (Day 1) or consumption of chocolate-, caffeine-, or xanthine-containing products within 48 hours prior to dosing (Day 1);
23. Consumption of substances known to induce or inhibit liver metabolic enzymes (including grapefruit, mango, dragon fruit, grapes or grape juice, oranges or orange juice that could affect drug absorption, distribution, metabolism, and excretion within 48 hours prior to dosing [Day 1]);
24. Participation in strenuous activity within 48 hours prior to dosing (Day 1);
25. Female subjects who are pregnant or breastfeeding, who have a positive serum or urine pregnancy test result, or who are unable or unwilling to take contraceptive or abstinence measures approved by the investigator during the study;
26. History of constipation or the inability to maintain regular bowel movements at least once a day for the subjects of Group C2 within 3 months before administration;
27. Considered unsuitable for inclusion in the study by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
The number, severity and type of adverse events, including changes in vital signs, physical examinations, laboratory safety tests and ECGs | 8 days max
  To evaluate the safety and tolerability of Aom0319 in healthy subjects

SECONDARY OUTCOMES:
Maximum plasma concentration in plasma (Cmax) | Day1-2 for SAD
  Pharmacokinetics
Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration in plasma (AUC0-t) | Day1-2 for SAD
  Pharmacokinetics
Area under the concentration-time curve extrapolated from time 0 to infinity in plasma (AUC0-∞) | Day1-2 for SAD
  Pharmacokinetics
AUC from time 0 to 12 hours (AUC0-12) | Day1-2
  Pharmacokinetics
AUC from time 0 to 24 hours (AUC0-24) | Day1-2
  Pharmacokinetics
Time of the maximum observed concentration in plasma (Tmax) | Day1-2 for SAD
  Pharmacokinetics
Terminal elimination half-life in plasma (t1/2) | Day1-2 for SAD
  Pharmacokinetics
Volume of distribution during the terminal phase in plasma (Vz) | Day1-2 for SAD
  Pharmacokinetics
Total clearance in plasma (CL) | Day1-2 for SAD
  Pharmacokinetics
Terminal elimination rate constant in plasma (λz) | Day1-2 for SAD
  Pharmacokinetics
Mean residence time in plasma (MRT) | Day1-2 for SAD
  Pharmacokinetics
Cumulative amount of dose recovered in urine from time 0 to 24 hours (Ae0-24) | Day1-2
  Urine and faeces for PK
Cumulative percentage of dose recovered in urine from time 0 to 24 hours (fe0-24) | Day1-2
  Urine and faeces for PK
Renal clearance in urine (CLr) | Day1-2
  Urine and faeces for PK

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Mclendon, PhD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No